CLINICAL TRIAL: NCT06770036
Title: Implementation Strategies for Caregiver and Teacher Use of Behavioral Interventions With ADHD: A Pilot Study, Aim 1
Brief Title: Caregiver Implementation Strategies Field Pre-Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-021965; R34MH132718-01A1 (NIH)
Record Dates: First submitted 2025-01-09; First posted 2025-01-13 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Attention Deficit Hyperactivity Disorder Symptoms
Keywords: Attention Deficit Hyperactivity Disorder; Positive Behavior Management; Inattentive; Hyperactive; Impulsive
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm; Impulsive Behavior | interventions — Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caregiver Resource Package (Experimental): Caregiver in this group will receive an implementation resource support package and will receive support in using it.
  Interventions: Behavioral: Implementation Resource Package for Caregivers

INTERVENTIONS:
Behavioral: Implementation Resource Package for Caregivers — The implementation resource package for caregivers is a set of resources provided to caregivers that aims to support their use of evidence-based behavior management practices and home-school communication strategies.
  Other Names: Supporting School Success - Caregiver Version; Positive Behavior Management Toolkit for Caregivers

SUMMARY:
The purpose of this study is to field pre-test an implementation strategy resource package that aims to support caregivers in using behavioral interventions for children with hyperactive, inattentive, or impulsive behaviors. Enrolled caregivers will be assigned to use the resource package with their children. The research team will collect quantitative and qualitative data regarding acceptability, appropriateness, and feasibility, in preparation for a randomized pilot study.

DETAILED DESCRIPTION:
Evidence-based interventions for children with or at-risk for Attention-Deficit/Hyperactivity Disorder (ADHD) include antecedent- and consequence- based behavioral interventions in both the classroom and home settings as well as effective home-school communication approaches. Schools are a promising setting in which to provide early intervention for mental health challenges and to increase access to mental health care. Furthermore, stronger integration between home- and school- based interventions has the potential to meaningfully improve child outcomes. However, there are substantial implementation challenges to caregivers' use of these evidence-based interventions. This study aims to field pre-test an implementation strategy resource package to support caregivers in using evidence-based behavioral interventions for children with hyperactive, inattentive, or impulsive behaviors. After an initial iterative process of developing the resource package, enrolled caregivers will use the resource package with their children in a single-arm study, for the purpose of assessing initial implementation outcomes and making final adjustments to the resource package.

ELIGIBILITY:
Inclusion Criteria:

* Students in or entering grades K-5 in the greater Philadelphia area
* Nominated for participation by a school staff member or parent/legal guardian
* Identified by that staff member or parent/legal guardian as displaying functional impairment from ADHD symptoms, as measured by a score of a 3 or greater on the modified version of the Impairment Rating Scale.

Exclusion Criteria:

* Presents as in acute risk of harm to self or others, such that participation in the study is clinically inappropriate because the child warrants more intensive intervention
* Special education classification of 'intellectual disability'
* Students from families in which there is not a caregiver who speaks English will be excluded because the focus of this study is developing an English-language version of the resource package

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-01-21 (Actual); Study Completion 2026-01-23 (Actual)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure | Endpoint (i.e, at least 8 weeks from resource package receipt)
  Caregiver-reported total score on the Feasibility of Intervention Measure (FIM), which consists of 4 items on a 5-point Likert scale (from 1 = Completely Disagree to 5 = Completely Agree). The total score is the average of the 4 item scores.
Acceptability of Intervention Measure | Endpoint (i.e, at least 8 weeks from resource package receipt)
  Caregiver -reported total score on the Acceptability of Intervention Measure (AIM), which consists of 4 items on a 5-point Likert scale (from 1 = Completely Disagree to 5 = Completely Agree). The total score is the average of the 4 item scores.
Intervention Appropriateness Measure | Endpoint (i.e, at least 8 weeks from resource package receipt)
  Caregiver -reported total score on the Intervention Appropriateness Measure (IAM), which consists of 4 items on a 5-point Likert scale (from 1 = Completely Disagree to 5 = Completely Agree). The total score is the average of the 4 item scores.
Change in observed caregiver fidelity to behavioral interventions | Baseline, Endpoint (i.e, at least 8 weeks from resource package receipt)
  A member of the study will conduct observations to measure fidelity of caregiver use of the behavioral interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn M Lawson, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided